CLINICAL TRIAL: NCT03022721
Title: Heidelberg Study on Diabetes and Complications
Acronym: HEIST-DiC
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Stefan Kopf MD, Head of the Clinical Study Center for Diabetes Research, Heidelberg University
Other Study IDs: S-383/2016
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Complications
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, PBMC, whole blood, urine. There is a possibility of DNA extraction from PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with diabetes: Patients with both type 1 and type 2 Diabetes will be enrolled, Independent of Diabetes Duration, therapy etc.
  No interventions are planned.
  Interventions: Other: No interventions are planned for this study.
- Pre-Diabetics: Patients who have either imparied fasting Glucose or impaired Glucose tolerance in the oral Glucose tolerance test.
  No interventions are planned.
  Interventions: Other: No interventions are planned for this study.
- Healthy controls: Study participants without Diabetes or Pre-diabetes in the oral Glucose tolerance test.
  no interventions are planned.
  Interventions: Other: No interventions are planned for this study.

INTERVENTIONS:
Other: No interventions are planned for this study. — No interventions are planned for this study, it is purely observational.

SUMMARY:
The prospective observational study entitled "Heidelberg Study on Diabetes and Complications" is designed to Monitor the presence and development of diabetic complications in type 1 and type 2 diabetic patients, as well as pre-diabetics. Mail Goal is to detect new metabolic mechanisms or new risk factors for the development of diabetic complications in order to identify risk-subgroups. Non-diabetic controls will be enrolled for reference and comparison.

DETAILED DESCRIPTION:
The prospective observational study entitled "Heidelberg Study on Diabetes and Complications" is designed to show that diabetes according to the current medical definition does not exist. Without question, there is an autoimmune disease that destroys beta cells in the pancreas, which leads to absolute insulin deficiency with consecutively elevated blood glucose levels. This disease is defined as diabetes mellitus type 1. Insulin treatment is absolutely necessary in this state, since absolute insulin deficiency leads to lipolysis with consecutive ketoacidosis and eventually death. On the other hand, type 2 diabetes is generally defined as relative insulin deficiency with consecutively elevated blood glucose levels. This disease is often mentioned in the context of the metabolic syndrome, which additionally comprises obesity, arterial hypertension, dyslipidemia, and cardiovascular diseases. Therefore, only the name "diabetes mellitus" is shared by these two diseases, which means "sweet flow", therefore only describing a symptom.

Multiple interventional studies were aimed on avoiding or reducing the development of late diabetic complications (nephropathy, neuropathy, retinopathy, microangiopathy). This is true for both type 1 and type 2 diabetes. Up to this day, no study was able to demonstrate that treatment of normalization of blood glucose levels reduces or even reverses development of these complications. Moreover, several type 2 diabetic patients developed typical diabetic complications before definitive manifestation of the actual disease.

Therefore, we hypothesize that late diabetic complications stand in no primary context with blood glucose control, but are associated with other metabolic disorders. One aspect are reactive metabolites (glyoxal, methylglyoxal, 3-DG), which are formed in glycolysis and lipolysis in the context of energy production of cells. These metabolites are detoxified to lactate by certain enzymes. In case this detoxification is compromised, or production of these metabolites elevated, so called advanced glycation endproducts (AGEs) can form. Moreover, within the process of energy production, reactive oxygen species (ROS) and oxydative stress are more pronounced, which can have direct influence on cellular metabolism. This interaction leads to inflammation and DNA damage. Survival of the cells is dependent on defense mechanisms, which seem to be genetically determined, with cellular ageing playing a role as well (cellular senescence). With advanced ageing, cells lose these defense mechanisms against these permanent metabolic attacks.

Therefore, the following hypotheses arise:

1. Diabetes mellitus type 2 is no independent disease, but a late complication of metabolic imbalance
2. Typical "late diabetic complications" are not based on insufficient blood glucose lowering therapy, but on the basis of this metabolic imbalance, and can therefore affect every patient, even without manifested "diabetes mellitus type 2"
3. Diabetes mellitus type 1 is an autoimmundisease with consecutive absolute insulin deficiency, however manifestation of late diabetic complications is based on the same metabolic dysbalance (overlap with type 2).

In order to investigate these hypotheses, study participants will be profoundly examined once yearly concerning glycemic metabolic state and clinical findings related to micro- and macrovascular diabetic complications, Moreover, reactive metabolites like AGEs, ROS, methylglyoxal, and DNA damage as well as other parameters associated with cellular senescence will be examined. We will also collect information concerning quality of life, well-being, depression, and neuropathic pain.

This is the first study of its kind to include non-diabetics, pre-diabetics, and diabetics with the possibility to study differences and common ground regarding cellular metabolism. Moreover, to the best of our knowledge, there is no precise clinical characterization of peripheral nerve function in pre-diabetics, although some of these patients already complain about neuropathic symptoms. In addition to that, the natural clinical course not only in diabetics, but also in pre-diabetics will be observed over a longer period of time. Finally, changes in surrogate markers over the natural course of pre-diabetes can be observed for the first time, onset of type 1 or type 2 diabetes can be registered immediately, and all patients can be directly compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria Age between 18 and 75 years Persons with manifest diabetes mellitus type 1 or type 2 and diagnosis according to DDG guidelines 2011, that is HbA1c of 6,5 percent or higher after exclusion of false values, more than 200 mg per dl two hours after glucose in the oGTT, fasting glucose more than 126 mg per dl, spontaneous glucose more than 200 mg per dl at least twice Healthy persons without diabetes or impairment of glucose metabolism in the oGTT according to DDG guidelines 2011 fasting plasma glucose less than 100 mg per dl and 2 hour plasma glucose less than 140 mg per dl Pre diabetics with impaired fasting glucose between 100 mg per dl and 125 mg per dl, or impaired glucose tolerance with 2 hour glucose values between 140 and 199 mg per dl in the oGTT, all values from venous plasma

Exclusion Criteria General exclusion criteria Secondary types of Diabetes, ADA criteria type 3 B H Current pregnancy Acute infections or fever Immune suppressant therapy Severe psychiatric diseases requiring treatment, including personality disorders, schizophrenia, depression Known alcohol or drug dependency Severe heart NYHA stadium IV, kidney, or liver insufficiency Non diabetic liver disease, for example PBC, PSC, Wilsons disease, hemochromatosis, autoimmune hepatitis severe peripheral artery disease stadium IV non diabetic glomerulopathy Cancer or other malignant diseases within the last 5 years Infectious diseases like hepatitis B, C, E, or HIV Other severe autoimmune diseases Current participation in an interventional study Anemia or disorders of bone marrow Exclusion criteria for MRI Pacemaker or ICD Metallic and magnetic implants, for example mechanic cardiac valves replacements, joint prostheses, clips after vascular surgery, middle or inner ear implants, recent tooth implants, penile implants Waist circumference more than 135 cm Claustrophobia Allergies against MRI contrast Impaired kidney function with a GFR less than 65 ml per min

Exclusion criteria for clamp study Past history of deep vein thrombosis or pulmonary embolism Routine laboratory test results less than 80 percent below lower reference value of Ferritin, iron, leucocytes, hemoglobin, hematocrite, RBC, platelets, blood alcohol Level

Exclusion criteria for bioimpedance measurement Pacemaker or ICD

Exclusion criteria for lung function testing Ignoring or non understanding of the instructions Body weight more than 160 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population comprises patients with Diabetes, patients with pre-diabetes, and healthy controls. In total, 500 participants shall be enrolled and observed for 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09; Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Development of diabetic complications | 10 years
  Diabetic complications include diabetic nephropathy, diabetic retinopathy, diabetic polyneuropathy, autonomous neuropathy, or macrovascular complications such as stroke, peripheral artery disease, or myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kopf, MD, Principal Investigator — Head of the Clinical Study Center for Diabetes Research
Locations (1):
- Department of Medicine, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data is planned.

REFERENCES:
- [Derived] Eldesouky O, Seebauer L, Rukwied R, Carr R, Roshan M, Gottlieb H, Tsilingiris D, Kopf S, Herzig S, Fleming T, Kessler J, Szendroedi J, Schmelz M, Kender Z. Mismatch between intact electrical excitability and lost heat pain in diabetic neuropathy. Pain. 2026 Jan 6. doi: 10.1097/j.pain.0000000000003898. Online ahead of print. PMID 41494160
- [Derived] Kliemank E, von Rauchhaupt E, Seebauer L, Roshan M, Ansmann M, Flegka V, Schimpfle L, Tsilingiris D, Bartl H, Fleming T, Kender Z, Jende JME, Mooshage CM, Schwarz D, Bendszus M, Schirmacher P, Herzig S, Nawroth PP, Kopf S, Szendroedi J, Sulaj A. Cohort profile of the Heidelberg study on diabetes and complications HEIST-DiC. Sci Rep. 2025 Aug 12;15(1):29580. doi: 10.1038/s41598-025-15343-8. PMID 40797027
- [Derived] Mooshage CM, Schimpfle L, Tsilingiris D, Kender Z, Aziz-Safaie T, Hohmann A, Szendroedi J, Nawroth P, Sturm V, Heiland S, Bendszus M, Kopf S, Jende JME, Kurz FT. Magnetization transfer ratio of the sciatic nerve differs between patients in type 1 and type 2 diabetes. Eur Radiol Exp. 2024 Jan 9;8(1):6. doi: 10.1186/s41747-023-00405-1. PMID 38191821
- [Derived] Mooshage CM, Tsilingiris D, Schimpfle L, Seebauer L, Eldesouky O, Aziz-Safaie T, Hohmann A, Herzig S, Szendroedi J, Nawroth P, Heiland S, Bendszus M, Kurz FT, Kopf S, Jende JME, Kender Z. A diminished sciatic nerve structural integrity is associated with distinct peripheral sensory phenotypes in individuals with type 2 diabetes. Diabetologia. 2024 Feb;67(2):275-289. doi: 10.1007/s00125-023-06050-y. Epub 2023 Nov 29. PMID 38019287
- [Derived] Mooshage CM, Tsilingiris D, Schimpfle L, Kender Z, Aziz-Safaie T, Hohmann A, Szendroedi J, Nawroth P, Sturm V, Heiland S, Bendszus M, Kopf S, Kurz FT, Jende JME. Insulin Resistance Is Associated With Reduced Capillary Permeability of Thigh Muscles in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e137-e144. doi: 10.1210/clinem/dgad481. PMID 37579325
- [Derived] Tsilingiris D, Schimpfle L, von Rauchhaupt E, Sulaj A, Seebauer L, Bartl H, Herzig S, Szendroedi J, Kopf S, Kender Z. Dysmetabolism-related Early Sensory Deficits and Their Relationship With Peripheral Neuropathy Development. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e979-e988. doi: 10.1210/clinem/dgad248. PMID 37139855
- [Derived] Jende JME, Groener JB, Kender Z, Hahn A, Morgenstern J, Heiland S, Nawroth PP, Bendszus M, Kopf S, Kurz FT. Troponin T Parallels Structural Nerve Damage in Type 2 Diabetes: A Cross-sectional Study Using Magnetic Resonance Neurography. Diabetes. 2020 Apr;69(4):713-723. doi: 10.2337/db19-1094. Epub 2020 Jan 23. PMID 31974140
- [Derived] Groener JB, Jende JME, Kurz FT, Kender Z, Treede RD, Schuh-Hofer S, Nawroth PP, Bendszus M, Kopf S. Understanding Diabetic Neuropathy-From Subclinical Nerve Lesions to Severe Nerve Fiber Deficits: A Cross-Sectional Study in Patients With Type 2 Diabetes and Healthy Control Subjects. Diabetes. 2020 Mar;69(3):436-447. doi: 10.2337/db19-0197. Epub 2019 Dec 11. PMID 31826867
- [Derived] Kopf S, Groener JB, Kender Z, Fleming T, Bischoff S, Jende J, Schumann C, Ries S, Bendszus M, Schuh-Hofer S, Treede RD, Nawroth PP. Deep phenotyping neuropathy: An underestimated complication in patients with pre-diabetes and type 2 diabetes associated with albuminuria. Diabetes Res Clin Pract. 2018 Dec;146:191-201. doi: 10.1016/j.diabres.2018.10.020. Epub 2018 Oct 31. PMID 30389624